CLINICAL TRIAL: NCT06916650
Title: Comparative Effectiveness of High-Intensity Laser Therapy Versus Corticosteroid Injection Versus Manual Therapy, Each Combined With Standard Exercise, for Frozen Shoulder (Adhesive Capsulitis): A Randomized Controlled Trial
Brief Title: Comparing HILT, Steroid Injection, and Manual Therapy for Frozen Shoulder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPARE-FS
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HILT + Standard Exercise (Experimental): Participants receive High-Intensity Laser Therapy (HILT) 2 times/week for 6 weeks, plus the Standard Exercise Program.
  Interventions: Device: High-Intensity Laser Therapy (HILT); Behavioral: Standard Exercise Program
- Corticosteroid Injection + Standard Exercise (Active Comparator): Participants receive a single ultrasound-guided intra-articular corticosteroid injection at baseline, plus the Standard Exercise Program.
  Interventions: Drug: Ultrasound-Guided Intra-articular Corticosteroid Injection; Behavioral: Standard Exercise Program
- Manual Therapy + Standard Exercise (Active Comparator): Participants receive manual therapy 2 times/week for 6 weeks, plus the Standard Exercise Program.
  Interventions: Behavioral: Manual Therapy; Behavioral: Standard Exercise Program
- Standard Exercise Alone (Active Comparator): Participants receive the Standard Exercise Program only.
  Interventions: Behavioral: Standard Exercise Program

INTERVENTIONS:
Device: High-Intensity Laser Therapy (HILT) — Nd:YAG laser (1064 nm) applied to anterior, lateral, posterior glenohumeral joint aspects. Three-phase protocol per session: (1) 10 J/cm² @ 10 Hz; (2) 12 J/cm² @ 2000 Hz; (3) 10 J/cm² @ 15 Hz. Total energy ~1200 J/session. Frequency: 2 sessions/week for 6 weeks (12 sessions total). Delivered by trained PTs.
  Arms: HILT + Standard Exercise
Drug: Ultrasound-Guided Intra-articular Corticosteroid Injection — Single injection into the glenohumeral joint under ultrasound guidance. Consists of 40 mg methylprednisolone acetate combined with 4 ml of 1% lidocaine hydrochloride. Delivered at baseline by an experienced orthopedic physician.
  Arms: Corticosteroid Injection + Standard Exercise
Behavioral: Manual Therapy — Skilled hands-on techniques including glenohumeral joint mobilizations (Maitland grades III-IV), posterior capsule stretching, scapular mobilization, and soft tissue techniques targeting restricted tissues. Session duration: ~30 minutes. Frequency: 2 sessions/week for 6 weeks (12 sessions total). Delivered by PTs specialized in manual therapy.
  Arms: Manual Therapy + Standard Exercise
Behavioral: Standard Exercise Program — Standardized program including pendulum exercises, active-assisted range of motion exercises (e.g., wand, wall climbs), stretching (e.g., cross-body, sleeper stretch), and progressive resistive exercises using resistance bands. Includes supervised instruction/progression and a daily home exercise program component. Supervised instruction frequency: 2 sessions/week for first 6 weeks, then 1 session/week for next 6 weeks (total 18 supervised sessions over 12 weeks). Delivered by trained PTs.

SUMMARY:
This study compares three common treatments for frozen shoulder when added to a standard exercise program: High-Intensity Laser Therapy (HILT), a corticosteroid (steroid) injection into the shoulder joint, and hands-on manual therapy by a physical therapist. A fourth group will receive only the standard exercise program. The goal is to see which combination works best to reduce shoulder pain and improve shoulder function over 6 months. The main outcomes are changes in pain (VAS scale) and shoulder disability (SPADI questionnaire) at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Age between 40 and 70 years, inclusive. Clinical diagnosis of primary (idiopathic) frozen shoulder, defined by shoulder pain and ≥50% restriction in passive external rotation compared to the contralateral (unaffected) shoulder.

Symptom duration between 3 and 9 months. Average shoulder pain intensity ≥ 4 on a 10-cm Visual Analogue Scale (VAS) over the past week.

Normal or age-appropriate radiographic findings of the glenohumeral joint (ruling out significant arthritis, fractures, calcific tendinitis).

Willingness and ability to attend scheduled treatment/assessment sessions. Ability to understand study procedures and provide written informed consent.

Exclusion Criteria:

Secondary frozen shoulder (e.g., post-traumatic, post-surgical, related to systemic disease like diabetes - clarify if diabetes is excluded or just secondary FS from diabetes).

Clinical or imaging evidence of significant rotator cuff tear requiring specific management.

Radiographic evidence of moderate to severe glenohumeral osteoarthritis (e.g., Kellgren-Lawrence grade ≥ 3).

Previous surgery on the index shoulder. Significant neurological disorders affecting shoulder or upper extremity function (e.g., cervical radiculopathy, stroke).

Received a corticosteroid injection in the index shoulder within the past 3 months.

Known contraindications to corticosteroid injections (e.g., uncontrolled diabetes, allergy, local infection).

Known contraindications to High-Intensity Laser Therapy (e.g., active malignancy in the treatment area, photosensitivity, pacemaker over treatment area).

Current participation in another interventional clinical trial for shoulder pain.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder Pain Intensity | Baseline (T0), 6 weeks (T1), 12 weeks (T2), 6 months (T3)
  Visual Analogue Scale (VAS) for Pain. Change from baseline in average shoulder pain over the past week, measured on a 10 cm horizontal VAS, where 0 cm = no pain and 10 cm = worst imaginable pain. Lower scores indicate less pain. MCID estimated at 1.4 cm.
Change in Shoulder Pain and Disability | Baseline (T0), 6 weeks (T1), 12 weeks (T2), 6 months (T3)
  Shoulder Pain and Disability Index (SPADI). Change from baseline in the total SPADI score. SPADI consists of 13 items assessing pain (5 items) and disability (8 items). Total score ranges from 0-100, with lower scores indicating less pain and disability.

SECONDARY OUTCOMES:
Change in Passive Shoulder Range of Motion (ROM) | Baseline (T0), 6 weeks (T1), 12 weeks (T2), 6 months (T3)
  Change from baseline in passive shoulder ROM measured in degrees for: External Rotation (at side), Abduction (in scapular plane), Flexion, and Internal Rotation (vertebral level reached). Measured using a standard goniometer.
Patient Global Rating of Change | 6 weeks (T1), 12 weeks (T2), 6 months (T3)
  Global Rating of Change (GRC) Scale. Patient's self-rated overall change in their shoulder condition since starting the study, measured on a Likert scale (e.g., 7-point scale from "very much worse" to "very much improved"). Assessed relative to baseline.
Incidence of Adverse Events | Throughout study participation (up to 6 months)
  Number, type, and severity of any adverse events (AEs) reported by participants or observed by study staff throughout the study duration, categorized by potential relationship to the assigned intervention (e.g., post-injection flare, skin reaction to HILT, increased pain after manual therapy/exercise).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No